CLINICAL TRIAL: NCT06740513
Title: The New Clinical Registration Trial of Interventional Treatment for Patients with Symptomatic Intracranial Artery Stenosis
Acronym: CRTICAS-2
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: CRTICAS-2
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Atherosclerotic Stenosis (ICAS); Stroke
Keywords: Intracranial atherosclerotic stenosis; clinical registration trial; interventional treatment; Medical Therapy plus Stent/Balloon Angioplasty; Endovascular Treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endovascular Treatment Group: all the participants in this group will be performed with endovascular treatment
  Interventions: Procedure: Endovascular Treatment

INTERVENTIONS:
Procedure: Endovascular Treatment — Medical Therapy plus Stent/Balloon Angioplasty

SUMMARY:
Background:

Intracranial atherosclerotic stenosis (ICAS) is a major etiology of stroke worldwide, especially in East and South Asia, accounting for up to 50% of all ischemic stroke. Previous three randomized clinical trials did not demonstrate the superiority of intracranial stenting over aggressive medical management for symptomatic intracranial atherosclerotic stenosis (sICAS). The SAMMPRIS and VISSIT trials demonstrated that aggressive medical management was superior to self-expanding stenting and balloon-expanding stenting for sICAS. The CASSISS trial showed no significant difference in the risk of stroke or death between self-expanding stenting and aggressive medical management for sICAS. But recent BASIS trial demonstrated that balloon angioplasty plus aggressive medical management, compared with aggressive medical management alone, lowered the risk of a composite outcome.

CRTICAS was a prospective, real-world registry with 26 participating centres. It demonstrated a lower complication rate in treating patients with symptomatic ICAS with endovascular therapy in a real-world context, compared with the preceding RCTs. Uneven development in endovascular technology, institutional experience and patient selection in different volumes of centres may have an impact on overall safety of this treatment. The patients were screened from December 2013 to December 2015, which was almost 10 years ago. In consideration of the development of imaging evaluation and interventional devices, the CRTICAS-2 aims to figure out the effect and safety of endovascular treatment plus medical management for sICAS patients nowadays.

Methods:

As a multicenter and prospective cohort study, it starts in December 2024, the observation is scheduled to be completed by December 2028, with a total of at least 1000 sICAS patients recruited. The information on clinical, radiological, and laboratory practices will be recorded objectively. All of the patients will be monitored until death or 12 months after the occurrence of symptomatic stroke.

Study Design:

In this study, an observational cohort will be set up. The primary outcome is the effect of endovascular treatment, which is subject to assessment using the total mortality and symptomatic stroke. The second outcome is the safety of endovascular treatment, with the postoperative ischemic complication. Based on the observation of the characteristics and outcome of sICAS patients, the ischemic events after surgery will be further addressed, and the function assessment system for operated sICAS patients will be established. We will detailedly collect the clinical data of all patients registered for the study includes medical record data; imaging examination; laboratory examination; hemodynamic evaluation and cognitive function evaluation. The imaging examination includes Magnetic Resonance Imaging(MRI), High-Resolution Magnetic Resonance Imaging(HRMRI), Computed Tomography Angiography(CTA), Magnetoencephalography (MEG) , Ultrasound and so on. The hemodynamic evaluation includes Optical CoherenceTomography (OCT), noninvasive FFR estimated from Phase Contrast Magnetic Resonance Angiography (PC-MRA) and so on. The cognitive function evaluation includes cognitive domains of verbal episodic memory, semantic verbal fluency, confrontation naming, mental processing speed-attention, executive function-cognitive flexibility and so on.

Objective:

To observe the effect of endovascular treatment plus medical therapy in patients with symptomatic intracranial atherosclerotic stenosis.

ELIGIBILITY:
Inclusion Criteria:

(1)18-80 years old; (2)Received endovascular therapy during hospitalization; (3) Intracranial arterial stenosis related to the following non-atherosclerotic factors will be not be considered: arterial dissection, moya-moya disease; vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebrospinal fluid pleocytosis; radiation-induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process, and suspected recanalized embolus; (4) Symptomatic intracranial stenosis: presented with transient ischemic stroke (TIA) or stroke within the past 12 months attributed to 70%-99% stenosis of a major intracranial artery (ICA, MCA [M1], vertebral artery, or basilar artery [BA]); (5) Degree of stenosis: 70%-99%; stenosis degree must be consistent with the criteria of endovascular treatment ; (6) No massive cerebral infarction (>1/2 MCA territory), intracranial hemorrhage, epidural or sub-dural hemorrhage, and intracranial brain tumor on CT or MRI scan; (7) Patient is willing and able to return for all follow-up visits required by the protocol; (8) Patient understands the purpose and requirements of the study, can make him/herself understood, and has signed informed consent.

Exclusion Criteria:

1. Patients had cerebrovascular diseases, e.g., intracranial aneurysm or vascular malformation, and intracranial tumors;
2. History of life-threatening allergy to contrast medium. If not life threatening and can be effectively pre-treated, patient can be enrolled at physicians' discretion;
3. Active bleeding diathesis or coagulopathy; active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets count <125,000, hematocrit <30, Hgb <10g/dL, uncorrected INR >1.5, bleeding time >1 minute beyond upper limit normal, or heparin-associated thrombocytopenia that increases the risk of bleeding, uncontrolled severe hypertension (systolic BP>180mmHg or diastolic BP>115mmHg), severe liver impairment (AST or ALT >3 times normal, cirrhosis), creatinine >265.2 mmol/L (unless on dialysis).
4. Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days or planned in the next 90 days after enrollment;
5. Severe dementia or psychiatric problems that prevent the patients from following an outpatient program reliably;
6. Pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All symptomatic intracranial atherosclerotic stenosis (sICAS) patients receiving endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of stroke or all-cause mortality | Within 30 days after surgery
  Stroke includes ischemic and hemorrhagic stroke, and is confirmed by postoperative imaging. Death defined as a mRS score of 6.
Stroke in the qualifying artery territory | After surgery 3 months, 6 months and 1 year.
  Including ischemic and hemorrhagic stroke, and confirmed by postoperative imaging.

SECONDARY OUTCOMES:
Changes of the National Institutes of Health Stroke Scale (NIHSS) score | After surgery 30 days, 3 months, 6 months, 1 year, 2 years and 3 years.
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit)
Changes in Modified Rankin Scale(mRS) | After surgery 3 months, 6 months and 1 year, 2 years and 3 years.
  The mRS score range from 0 (no disability) to 6 (death)
Stroke in the qualifying artery territory | After surgery 2 years and 3 years.
  Including ischemic and hemorrhagic stroke, and confirmed by postoperative imaging.
All-cause mortality | After surgery 1 year, 2 years and 3 years.
  Death defined as a mRS score of 6
Cognitive assessment score | After surgery 3 months, 6 months and 1 year, 2 years and 3 years.
  The cognitive function evaluation includes cognitive domains of verbal episodic memory, semantic verbal fluency, confrontation naming, mental processing speed-attention, executive function-cognitive flexibility and so on.
Serious Adverse Event | After surgery 30days, 3 months, 6 months and 1 year, 2 years and 3 years.
  Myocardial infarction, epilepsy and any adverse events requiring unexpected surgical treatment.
EQ-5D-5L | After surgery 1 year, 2 years and 3 years.
  The EQ-5D 5-Levels (EQ-5D-5L) range from 5 (no problems) to 25 (extreme problems), which deceased patients have a utility of 0.
Self-Rating Depression Scale(SDS) or Hamilton Depression Scale(HDRS) | After surgery 1 year, 2 years and 3 years.
  SDS range from 25 (Normal) to 100 (Very Severe Depression); HDRS range from 0 (Normal) to 42 (Very Severe Depression).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China